CLINICAL TRIAL: NCT04399447
Title: The Multi-center Normal Reference Study of Tissue Motion Tracking of Mitral Annular Displacement(TMAD) in Chinese Han Adults Study
Brief Title: Multicenter Normal Reference Study of Tissue Motion Tracking of Mitral Annular Displacement(TMAD)
Acronym: TMAD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Weidong Ren (Other)
Responsible Party: Sponsor-Investigator, Weidong Ren, Chief of Ultrasound, Shengjing Hospital
Organization: Shengjing Hospital (Other)
Other Study IDs: ShengJing Hospital Ultrasound
Record Dates: First submitted 2020-05-09; First posted 2020-05-22 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Left Ventricular Systolic Dysfunction; Healthy Volunteers
Keywords: systolic function; left ventricular; normal
MeSH Terms: conditions — Ventricular Dysfunction, Left

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- 18-29 year-old group: Based on the inclusion crtiteria, 200 healthy Han people at aged 18-29 and both sexes will be recruited in the analysis. Normal reference values of tissue motion tracking of mitral annular displacement will be obtained.
  Interventions: Radiation: Echocardiography
- 30-39 year-old group: Based on the inclusion crtiteria, 200 healthy Han people at aged 30-39 and both sexes will be recruited in the analysis. Normal reference values of tissue motion tracking of mitral annular displacement will be obtained.
  Interventions: Radiation: Echocardiography
- 40-49 year-old group: Based on the inclusion crtiteria, 200 healthy Han people at aged 40-49 and both sexes will be recruited in the analysis. Normal reference values of tissue motion tracking of mitral annular displacement will be obtained.
  Interventions: Radiation: Echocardiography
- 50-59 year-old group: Based on the inclusion crtiteria, 200 healthy Han people at aged 50-59 and both sexes will be recruited in the analysis. Normal reference values of tissue motion tracking of mitral annular displacement will be obtained.
  Interventions: Radiation: Echocardiography
- 60-69 year-old group: Based on the inclusion crtiteria, 200 healthy Han people at aged 60-69 and both sexes will be recruited in the analysis. Normal reference values of tissue motion tracking of mitral annular displacement will be obtained.
  Interventions: Radiation: Echocardiography
- 70-79 year-old group: Based on the inclusion crtiteria, 200 healthy Han people at aged 70-79 and both sexes will be recruited in the analysis. Normal reference values of tissue motion tracking of mitral annular displacement will be obtained.
  Interventions: Radiation: Echocardiography

INTERVENTIONS:
Radiation: Echocardiography — left ventricular systolic function of all participants were measured by tissue motion tracking of mitral annular displacement using PHILIPS

SUMMARY:
To establish the range of TMADmid、TMADmidpt% by using tissue motion tracking of mitral annular displacement (TMAD), and to explore the influencing factors.

DETAILED DESCRIPTION:
With the gradual aging of Chinese population and continuous development of economy and society, the incidence of cardiovascular disease and the number of patients have increased rapidly. The National Heart Center has reported that the number of patients with clinically diagnosed cardiovascular disease in China has reached 290 million in 2016 (240 million in 2014). Cardiovascular disease is the most common cause of death in humans. Left ventricular systolic function plays an important role in the treatment and prognosis of patients with myocardial diseases. Early sensitive detection of left ventricular systolic function, timely treatment and early evaluation of the therapeutic effect can greatly reduce the death of patients with myocardial diseases rate.

At present, the left ventricular ejection fraction (LVEF), measured by the two-plane Simpson method in clinical, is one of the methods to evaluating left ventricular systolic function. It is especially suitable for patients with geometric deformation of the left ventricle, but some early heart failure patients' LVEF is still in the normal range, whose systolic function has been reduced, but. In recent years, 2D longitudinal strain is one of the indicators for evaluating left ventricular systolic function. The researchers believe that 70% of cardiac function is obtained by longitudinal movement of myocardium , which can be used as a good indicator for identifying myocardial diseases. However, both the two-plane Simpson method and the 2D longitudinal strain require good sound transmission conditions and good image quality. You can clearly see the endocardium and epicardium. Not all of patients in the clinic can get better image.

Basic and clinical studies and clinical statistics show that tissue motion tracking of mitral annular displacement (TMAD) is not affected by image quality and can effectively evaluate left ventricular systolic function. It can measure the mitral valve annulus displacement by marking the mitral valve annulus point and the reference point, which can quickly and accurately evaluate the left ventricular longitudinal contraction function.

ELIGIBILITY:
Inclusion Criteria:

1. Han nationality
2. Ages 18-79.
3. Normal body mass index (18-25kg / m2).
4. Normal blood pressure (139-90 / 89-60mmHg).
5. No history of cardiovascular and respiratory diseases.
6. No abnormality was found in physical examination of cardiovascular and respiratory system.
7. Blood glucose, lipid profile and electrocardiogram were normal.
8. Echocardiography showed no structural heart disease and normal heart function.
9. No history of medications affecting cardiovascular system.

Exclusion Criteria:

1. Clinically significant or moderate heart valve regurgitation.
2. Respiratory diseases: acute or chronic respiratory diseases.
3. Endocrine diseases: thyroid disease, diabetes, hyperaldosteronism, pheochromocytoma, and abnormal adrenal function.
4. Anemia.
5. Pregnant or lactating women.
6. Abnormal liver function (glutamyl aminotransferase exceeds 2.0 times the upper limit of normal value), abnormal renal function (creatinine exceeds the normal value), increased blood lipids (triglycerides, total cholesterol, low density and high density lipoprotein, any of which is higher than Normal value).
7. Connective tissue disease.
8. Tumor.
9. Aortic and peripheral vascular diseases: aortic dilatation, aortic dissection, aortic constriction, multiple arteritis, and atherosclerosis.
10. Drink more than 50ml of white wine daily; more than 100ml of red wine; more than 300ml of beer.
11. Professional athletes.
12. The poor quality of the ultrasound image cannot satisfy the parameter measurement and analysis.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 2400 healthy adults with normal physical examination items will be selected from the physical examination center. According to sex and age stratification, totally 2400 cases will contain 1200 males and 1200 females. From 18 to 79 years old, they will be divided into 6 groups: 18-29 years, 30-39 years, 40-49 years, 50-59 years, 60-69 years and 70-79 years (n=400 per group).
Sampling Method: Probability Sample
Enrollment: 2400 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
left ventricular systolic function was measured by tissue motion tracking of mitral annular displacement（TMAD） | 1 day
  To establish the range of TMADmid by using TMAD
left ventricular systolic function was measured by tissue motion tracking of mitral annular displacement（TMAD） | 1 day
  To establish the range of TMADmidpt% by using TMAD

SECONDARY OUTCOMES:
left ventricular systolic function was measured by the two-plane Simpson method | 1 day
  the left ventricular ejection fraction measured by the two-plane Simpson method, is the standard of the clinical

OTHER OUTCOMES:
Serum biochemical index | 1 day
  Serum laboratory testing for blood cholesterol level (total cholesterol, HDL (high-density lipoprotein), LDL (low-density lipoproteins), triglycerides), fasting blood-glucose will be examed.

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Ren, Principal Investigator — Shengjing Hospital of China Medical Univeristy
Locations (75):
- China (75):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Gansu Baiyin Second People's Hospital, Baiyin, Gansu
  - The First People's Hospital of Foshan City, Foshan, Guangdong
  - The People's Hospital of Gaozhou, Gaozhou, Guangdong
  - the Second Affiliated Hospital of Guangzhou University of Chinese Medicine, Guangzhou, Guangdong
  - Qingyuan People's Hospital, Qingyuan, Guangdong
  - Affiliated Hospital of YouJiang Medical University for Nationalities, Baise City, Guangxi
  - People'S Hospital of Baise, Baise City, Guangxi
  - The People'S Hospital of Chong Zuo, Chongzuo, Guangxi
  - Guigang City People'S Hospital, Guigang, Guangxi
  - Laibin People's Hospital, Laibin, Guangxi
  - Guangxi International Zhuang Medical Hospital, Nanning, Guangxi
  - Guangxi Minzu Hospital, Nanning, Guangxi
  - The first peopel's hospital of yulin, Yulin, Guangxi
  - The First Affiliated Hospital of Hainan Medical University, Haikou, Hainan
  - Nanyang Second People's Hospital, Nanyang, He'nan
  - Fengning Manchu Autonomous County Hospital, Chengde, Hebei
  - Handan First Hospital, Handan, Hebei
  - shijiazhuang No.1 Hospital, Shijiazhuang, Hebei
  - The Fourth Hospital of Heibei Medical University Hebei Cancer Hospital, Shijiazhuang, Hebei
  - Tangshan fengnan district hospital, Tangshan, Hebei
  - Xingtai Third Hospital, Xingtai, Hebei
  - Mudanjiang Cardiovascular Hospital, Mudanjiang, Heilongjiang
  - The Third Affiliated Hospital of Qiqihar Medical Hospital, Qiqihar, Heilongjiang
  - People'S Hospital of Hunan Province, Changsha, Hunan
  - The First People's Hospital of Huaihua, Huaihua, Hunan
  - The First Affiliated Hospital of Baotou Medical College, Baotou, Inner Mongolia
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - Jiujiang University Affiliated Hospital, Jiujiang, Jiangxi
  - Baicheng Central Hospital, Baicheng, Jilin
  - Jilin Central General Hospital, Jilin, Jilin
  - Benxi Central Hospital, Benxi, Liaoning
  - Chaoyang Central Hospital, Chaoyang, Liaoning
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Dalian Municipal Central Hospital, Dalian, Liaoning
  - The Second Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - DanDong central hospital, Dandong, Liaoning
  - Fuchun Central Hospital, Fushun, Liaoning
  - General Hospital of Fushun Mining Bureau, Fushun, Liaoning
  - The First Affiliated Hospital of Jinzhou Medical University, Jinzhou, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Central Hospital Affiliated To ShenYang Medical College, Shenyang, Liaoning
  - The First Affiliated Hospital of Liaoning University of Traditional Chinese Medicine, Shenyang, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - The People'S Hospital of Liaoning Province, Shenyang, Liaoning
  - the Second Affiliated Hospital Of Shenyang Medical College, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Qinghai Provincial People's Hospital, Xining, Qinghai
  - The Second Hospital of Shandong University, Jinan, Shandong
  - Liaocheng People'S Hospital, Liaocheng, Shandong
  - Yantai Affiliated Hospital of Binzhou Medical University, Yantai, Shandong
  - Zibo City Linzi District People's Hospital, Zibo, Shandong
  - Shanghai Pudong New District Zhoupu Hospital, Shanghai, Shanghai Municipality
  - Baoji Central Hospital, Baoji, Shanxi
  - Hanzhong Central Hospital, Hanzhong, Shanxi
  - Xianyang Central Hospital, Xianyang, Shanxi
  - Shaanxi Provincial People'S Hospital, Xi’an, Shanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Affiliated Hospital of Chengdu University of Traditional Chinese Medicine, Chengdu, Sichuan
  - Chengdu First People's Hospital, Chengdu, Sichuan
  - Chengdu Second People'S Hospital, Chengdu, Sichuan
  - Chengdu Third People's Hospital, Chengdu, Sichuan
  - The Peoplep'S Hospital of Wenjiang District,Chengdu, Chengdu, Sichuan
  - West China-Guang'An Hospital,Sichuan University, Guang’an, Sichuan
  - The People's Hospital Of Leshan, Leshan, Sichuan
  - The Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan
  - Affiliated Hospital of North Sichuan Medical College, Nanchong, Sichuan
  - Nanchong Central Hospital, Nanchong, Sichuan
  - Panzhihua Central Hospital, Panzhihua, Sichuan
  - Suining Central Hospital, Suining, Sichuan
  - First Affiliated Hospital,School of Medical,Shihezi University, Shihezi, Xinjiang
  - Urumqi Friendship Hospital, Ürümqi, Xinjiang
  - Dali Bai Autonomous Prefecture People'S Hospital, Dali, Yunnan

IPD SHARING:
Plan to Share IPD: Undecided